CLINICAL TRIAL: NCT06174025
Title: Validity and Reliability of the 6 Minute Pegboard Ring Test in Duchenne Muscular Dystrophy Patients
Brief Title: Validity and Reliability of the 6 Minute Pegboard Ring Test
Status: Completed | Type: Observational
Sponsor: Çağtay Maden (Other)
Responsible Party: Sponsor-Investigator, Çağtay Maden, Assistant professor, Gaziantep Islam Science and Technology University
Organization: Gaziantep Islam Science and Technology University (Other)
Other Study IDs: 2023/236
Record Dates: First submitted 2023-11-20; First posted 2023-12-18 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; 6 Minute Pegboard and Ring Test; arm exercise endurance; upper extremity
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to investigate the validity and reliability of 6PBRT in individuals with DMD and its applicability on these patients.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is the most common type of progressive muscular dystrophies and is an X-linked recessive, rarely autosomal dominant, muscle disease. DMD begins in childhood and progresses until they become unable to walk. Individuals with DMD experience skeletal muscle weakness, difficulty breathing, and decreased exercise capacity. In these patients, traditionally lower extremity tests are; 6-minute walk tests, treadmill tests and Cardiopulmonary exercise tests are used. However, it is reported that the upper extremity is also affected in individuals with DMD. The 6-Minute Pegboard and Ring Test (6PBRT), which is valid and reliable in most disease groups, is also a test that can be applied to the upper extremities. It is important to use 6PBRT frequently in clinical research practice for patients with DMD and to know its validity and reliability. To our knowledge, the validity and reliability of this test in individuals with DMD has not been established in the literature. This study aimed to investigate the validity and reliability of 6PBRT in individuals with DMD and its applicability on these patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being diagnosed with Duchenne muscular dystrophy between the ages of 6-17,
* Being Level 1 and 2 according to the Brooke Upper Extremity Functional Classification Scale
* Having no problems reading and/or understanding the scales and cooperating with the tests to be.
* Ability to sit independently for approximately 15 minutes during the evaluation

Exclusion Criteria:

* Not volunteering to participate in the research,
* Having any orthopedic problem in the upper extremity,
* A neurological disease or other clinical condition that may affect cognitive status having a diagnosis,
* Having had surgery on the upper extremities in the last 6 months and any having an injury
* At a level that prevents functional activities in the upper extremity Having severe contractures (joint restriction)

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals diagnosed with Duchenne muscular dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
6 Minute Pegboard and Ring Test | A total of two measurements will be made at 1-week intervals within 6 months.
  The 6-minute pegboard and ring test is used to assess upper extremity functional capacity. The patient sat in front of a perforated board with bottom pegs at shoulder level. The upper pegs are placed in the hole 20 cm above the lower pegs. 10 rings of the same size are placed on the lower pegs. The patient is asked to move as many rings as possible from the lower pegs to the upper pegs and vice versa within a 6-minute period. Pulse, blood pressure, SpO₂, dyspnea and arm fatigue detection are recorded before/after each test. Before the actual test, patients are allowed to move up and down the rings in a cycle to become familiar with the testing procedure. If the patient wants to rest during the test, he is allowed, but the stopwatch is not stopped. During the test, standard encouraging phrases are said to the patient at the end of each minute.

SECONDARY OUTCOMES:
Quick Shoulder-Hand Syndromes Questionnaire | A total of two measurements will be made at 1-week intervals within 6 months.
  The Quick Shoulder-Hand Syndromes Questionnaire is used to evaluate musculoskeletal physical function and symptoms of the upper extremity. The survey consists of 11 items and is scored between 0-100 points. Higher scores indicate more disability
Assessment of muscle strength | A total of two measurements will be made at 1-week intervals within 6 months.
  Muscle strength will be measured using a digital dynamometer (Manual Muscle Tester™), shoulder flexor, shoulder abductor, elbow extensor and elbow flexor muscle strength. Muscle tests will be repeated three times for each side and the highest value will be recorded in kg. Muscle strength will be calculated as percentages of expected values.
The Pediatric Quality of Life Inventory | A total of two measurements will be made at 1-week intervals within 6 months.
  The health-related quality of life of the participants will be evaluated with the Turkish version PedsQL-3.0 Neuromuscular Module. The scale consists of 3 categories containing 25 items. These categories; It includes 17 items regarding the disease process and related symptoms, 3 items regarding communication skills, and 5 items regarding the family's financial and social support systems. The items of the scale are scored between 4 (always poses a problem) and 0 (never poses a problem). At the end of the scale, a score between 0 and 4 is made. A score close to 100 indicates that the health-related quality of life is at a better level.
Brooke Upper Extremity Functional Classification Scale | A total of two measurements will be made at 1-week intervals within 6 months.
  It will be used to evaluate the upper extremity functional level of the individuals who will be included in the study. It was developed to determine the functional level of the upper extremity in the clinical evaluation of DMD (11). The steps of this scale are as follows; Level 1: Begins to move with the arms at the sides and can fully clasp the hands above the head.
  Level 2: However, he can bring his arms above his head by flexing his elbows or use his accessory muscles Level 3: He cannot raise his hands above his head, but he can bring the glass to his mouth (uses both hands if necessary).
  Level 4: He can raise his hands to his mouth, but cannot lift a glass of water to his mouth.
  Level 5: Cannot raise hands to mouth, but can raise hands to hold a pen or pick up a coin from the table.
  Level 6: He cannot raise his hands up to his mouth and cannot use his hands functionally.

CONTACTS AND LOCATIONS:
Overall Officials: Çağtay MADEN, PhD, Principal Investigator — Gaziantep İslamic Science and Technology University
Locations (1):
- Gaziantep İslamic Science and Technology University, Gaziantep, Şahinbey, Turkey (Türkiye)

REFERENCES:
- [Derived] Maden C, Karabulut DG, Yigit S. Validity and Reliability of the 6-min Pegboard and Ring Test in Patients With Duchenne Muscular Dystrophy. Muscle Nerve. 2025 Feb;71(2):200-207. doi: 10.1002/mus.28314. Epub 2024 Dec 11. PMID 39660725